CLINICAL TRIAL: NCT03496142
Title: Perineal Versus Rectal Approach for Prostate Biopsy to Prevent Iatrogenic Infections
Acronym: PRAPI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institut Mutualiste Montsouris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: URO-03-2017
Record Dates: First submitted 2018-04-05; First posted 2018-04-12 (Actual); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Prostate Cancer
Keywords: Prostate biopsy approach; Transrectal prostate biopsy; Transperineal prostate biopsy; Iatrogenic infection; Prevention
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients who will have prostate biopsy will be randomized 1:1 among transperineal or transrecal approach
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transperineal prostate biopsy (Active Comparator): Patient will have a transperineal prostate biopsy.
  Interventions: Procedure: Transperineal prostate biopsy
- Transrectal prostate biopsy (Active Comparator): Patient will have a transrectal prostate biopsy.
  Interventions: Procedure: Transrectal prostate biopsy

INTERVENTIONS:
Procedure: Transperineal prostate biopsy — Puncture of 12 to 30 percutaneous prostate core biopsies through the perineum with a transrectal ultrasound probe guidance. The procedure would be performed with the Artemis (Eigen) device allowing topographic recording of the puncture and MRI / ultrasound image fusion in order to target the MRI suspected lesion.
  Arms: Transperineal prostate biopsy
Procedure: Transrectal prostate biopsy — Patient would undergo 12 to 30 transrectal prostate core biopsies through the rectum with a transrectal ultrasound probe guidance. The procedure would be performed with the Artemis (Eigen) device allowing topographic recording of the puncture and MRI / ultrasound image fusion in order to target the MRI suspected lesion.
  Arms: Transrectal prostate biopsy

SUMMARY:
Retrospective reports from literature have shown a lower rate of infections for transperineal versus transrectal approach for prostate biopsies in the setting of prostate cancer suspicion.

The aim of this study would be to compare in a prospective randomized trial the rate of infection with transperineal versus transrectal approach.

DETAILED DESCRIPTION:
Retrospective reports from literature have shown a lower rate of infections for the transperineal versus transrectal approach for prostate biopsies in the setting of prostate cancer suspicion.

Post-biopsy infection is becoming a more and more challenging situation due to the increase of incidence and development of antibiotic resistant germs.

The aim of this study would be to compare in a prospective randomized trial the rate of infection with transperineal vs transrectal approach.

Patient presenting an indication of prostate biopsy (PSA elevation, suspicious lesion at digital rectal, suspicious lesion on MRI) would be randomized 1:1 among transrectal vs transperineal biopsies.

Post-biopsy infection would be monitored by systemic urine analysis at one, two and four weeks after procedure and in case of clinical symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Indication of prostate biopsy

Exclusion Criteria:

* No indication of prostate biopsy
* Impossibility for prostate biopsy (e.g. major anal stenosis or history of anal amputation)
* Antibiotic treatment within three months before prostate biopsy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2018-04 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Rate of post-biopsy infection from Baseline to four weeks after prostate biopsy | Four weeks post-biopsy
  Urinary infection will be assessed based on urinanalysis : 10^5 germs and 10^4 leucocytes minimum)

SECONDARY OUTCOMES:
Presence of antibiotic resistant germ | One week, two weeks and four weeks post-biopsy
  Antibiotic resistant germ will be assessed on urinanalysis
Presence of complication post-biopsy : hematuria, urinary retention, rectoragy, any other complication | One week, two weeks and four weeks post-biopsy
  Presence of complication will be assessed during phone interview with the patient

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre INGELS, MD, Principal Investigator — Institut Mutualiste Montsouris
Locations (1):
- Institut Mutualiste Montsouris, Paris, France

IPD SHARING:
Plan to Share IPD: No